CLINICAL TRIAL: NCT06422013
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-design Clinical Study to Evaluate the Body Fat Reducing Effect and Safety of Lactiplantibacillus Plantarum APsulloc 331261(GTB1)
Brief Title: Clinical Study to Evaluate the Body Fat Reducing Effect and Safety of GTB1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amorepacific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AP-PV-2022-01
Record Dates: First submitted 2024-05-15; First posted 2024-05-20 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Body Fat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GTB1 (Active Comparator): Once-daily, once a packet, for 12 week
  Interventions: Dietary Supplement: GTB1
- Placebo (Placebo Comparator): Once-daily, once a packet, for 12 week
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: GTB1 — oral administration of GTB1 powder packet once daily
  Arms: GTB1
Dietary Supplement: Placebo — oral administration of placebo powder packet once daily
  Arms: Placebo

SUMMARY:
This study was conducted to investigate the effects of daily supplementation of GTB1 on decrease of body fat.

DETAILED DESCRIPTION:
This study was a 12 week, randomized, double-blind, placebo-controlled human trial. 100 subjects were randomly divided into GTB1 group and placebo group. It is to evaluate the changes in the displayed evaluation items when taking GTB1 once a day, in comparison with taking a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged between 19~65 years at the screening
* Participants who were BMI 25.0~34.9 kg/m^2 (Excluding those who need to take or be prescribed medication that affects fat reduction, if the BMI is between 30.0~34.9 kg/m^2)
* Participants who have a waist circumference of 90 cm for men and 85 cm or more for women
* Participants who have fully understood the information provided about the study voluntarily decided to participate and agreed to comply with precautions

Exclusion Criteria:

* Participants who decrease 10% more of weight within 3 months period to the screening
* Participants who have undergone surgical procedures (such as gastrectomy) for weight loss
* Participants who have a history of malignant tumors within 5 years prior to participating in the clinical study
* Participants who have a systolic blood pressure of 160 mmHg or higher, or a diastolic blood pressure of 100 mmHg or higher (those who are stably controlling their blood pressure with medication can participate)
* Participants who are taking beta-blockers or diuretics as part of their hypertension treatment
* Patients who have been diagnosed with Type 1 or Type 2 diabetes and are taking oral hypoglycemic agents and insulin
* Participants who have taken antibiotics within 4 weeks prior to the screening examination
* Participants who have taken health functional foods, herbal medicine, or general foods for the purpose of weight loss within 4 weeks prior to the screening visit
* Participants with clinically significant acute or chronic diseases of the cardiovascular system, endocrine system, immune system, respiratory system, liver biliary system, kidney and urinary system, neuropsychiatry system, musculoskeletal system, inflammatory and hematologic, gastrointestinal diseases, and other diseases requiring treatment
* Participants with a past history of gastrointestinal diseases (e.g., Crohn's disease) or gastrointestinal surgery (but, excluding simple cecal surgery and hernia surgery) that can affect the absorption of products of the human trial
* Participants who have participated in other clinical study within 3 months prior to the screening examination
* Women who are pregnant or breastfeeding
* Women who may become pregnant and have not used appropriate contraceptives
* Participants who show the following relevant results in a Laboratory test

  * Aspartate Transaminase (AST), Alanine Transaminase (ALT) > Reference range 3 times upper limit
  * Serum Creatinine > 2.0 mg/dl
* Participants who the principal investigator judged inappropriate for the participant in this study because of a laboratory test result, etc.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
Changes of percent body fat(trunk, total ect.) | Baseline, Week 12
  Measurement is made using dual-energy X-ray absorptiometry(DEXA)

SECONDARY OUTCOMES:
Changes of fat free mass(trunk, total ect.) | Baseline, Week 12
  Measurement of the target area is made using dual-energy X-ray absorptiometry (DEXA)
Changes of total abdominal fat area, visceral fat area and subcutaneous fat area | Baseline, Week 12
  Measurement of the target area is made using computed tomography (CT)
Changes of waist, hip circumference and waist/hip circumference ratio | Baseline, Week 12
  Measurement of waist and hip circumference is performed following the WHO guideline
Changes of indicator of lipid metabolism | Baseline, Week 12
  Indicator of lipid metabolism(i.e., Total cholesterol, Triglyceride, LDL-cholesterol, HDL-cholesterol)
Changes of obesity-related hormone index | Baseline, Week 12
  Obesity-related hormone indexes(Adiponectin, Leptin etc.). As blood adiponectin levels increase, blood leptin concentrations decrease, indicating a positive change.

CONTACTS AND LOCATIONS:
Locations (1):
- Jeonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea

IPD SHARING:
Plan to Share IPD: No